CLINICAL TRIAL: NCT02582164
Title: Long-Working Distance OCT System With Fixation Alignment for Pediatric Imaging
Brief Title: Long-Working Distance OCT for Children
Acronym: LWDOCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Johns Hopkins University (Other); The Hartwell Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00060018
Record Dates: First submitted 2015-09-03; First posted 2015-10-21 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Retinal Diseases; Optic Nerve Diseases
Keywords: Optical Coherence Tomography (OCT); Swept Source OCT
MeSH Terms: conditions — Retinal Diseases; Optic Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Adult (Experimental): Duke Biomedical Engineering's long-working distance OCT system imaging of adult participants ages ≥18 year of age
  Interventions: Device: Duke Biomedical Engineering's Long-working distance OCT
- Teenage minors (Experimental): Duke Biomedical Engineering's long-working distance OCT system imaging of children ≥13-≤17 years of age
  Interventions: Device: Duke Biomedical Engineering's Long-working distance OCT
- Children-pre teen (Experimental): Duke Biomedical Engineering's long-working distance OCT system imaging of children ≥7-≤12 years of age
  Interventions: Device: Duke Biomedical Engineering's Long-working distance OCT
- Target age group ≥6 months to ≤6 years (Experimental): Duke Biomedical Engineering's long-working distance OCT system imaging of children ≥6 months to ≤6 years of age
  Interventions: Device: Duke Biomedical Engineering's Long-working distance OCT

INTERVENTIONS:
Device: Duke Biomedical Engineering's Long-working distance OCT — The long-distance SSOCT system designed by Duke University Biomedical Engineering Department allows the user to quickly image an eye at a much greater distance (typically 20-40 cm away but this could be longer or shorter). This could potentially be used while briefly attracting a child's attention to an illuminated image over the imaging lens. With this methodology, young patients would not need to place their eye close to the system and could be rapidly imaged during the short interval while they glance at the image from the correct distance.
  Other Names: LWD OCT

SUMMARY:
Young children age 6 month to 6 years are often not able to cooperate for advanced OCT eye imaging. The purpose of this study is to investigate the use of a novel long-working distance swept source (SS) optical coherence tomography imaging system with fixation alignment for use first in young adults, older children, and then young children ages 6 months to 6 years. The investigator's future goal is to obtain important retinal and optic nerve information from OCT in clinic in these young children.

DETAILED DESCRIPTION:
The overall objective of this study is to examine the utility of a long-working distance high speed SSOCT system along with technology to identify and use movies, etc. to aid with fixation. This study would be the first testing of such a system, first in adults and then moving to older children who could provide feedback, and then to young children.

This imaging data will be compared to other clinical tests and images collected during regular health care and eye examinations.

ELIGIBILITY:
Inclusion Criteria:

* Minor or adult undergoing eye examination at Duke Eye Center
* Adults with normal eye health enrolled as controls

Exclusion Criteria:

* Have any ocular disease that restricts the ability to perform OCT scanning
* Minor under the age of 6 months

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-06; Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Percent of eyes with successful research imaging. | 1 year
  The primary outcome of this study is the percent of eyes with successful research imaging of retinal and optic nerve microanatomy including the following: the inner surface and retinal pigment epithelial (RPE) layers of the macula, a full cross section of optic nerve, identification of either foveal center or severe pathology that obscures foveal depression and the presence or absence of 5 substructures of retina (Inner retinal complex, inner nuclear layer, outer plexiform layer, photoreceptor layer, RPE layer).

SECONDARY OUTCOMES:
Percent of eyes with 5 substructures of retina capable of being determined as deformed, containing cystoid spaces or abnormal (> 50%) thickening or thinning of layers. | 1 year
  Evaluation of retinal substructure morphology. Five substructures of retina include: Inner retinal complex, inner nuclear layer, outer plexiform layer, photoreceptor layer, RPE layer.
Participant feedback, as measured by questionnaire. | 1 year
  Scoring of participant feedback from questionnaire on: longevity of imaging, ease of finding or fixating on a target and comfortability during imaging. Parents and children will complete questionnaire together.
The time it takes to gather the research images. | 1 year
  The time from start of attempted imaging to imaging of both the macula and optic nerve of each eye.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Toth, MD, Principal Investigator — Duke University Health System, Department of Ophthalmology
Locations (1):
- Duke Eye Center, Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- [Background] Rothman AL, Tran-Viet D, Gustafson KE, Goldstein RF, Maguire MG, Tai V, Sarin N, Tong AY, Huang J, Kupper L, Cotten CM, Freedman SF, Toth CA. Poorer neurodevelopmental outcomes associated with cystoid macular edema identified in preterm infants in the intensive care nursery. Ophthalmology. 2015 Mar;122(3):610-9. doi: 10.1016/j.ophtha.2014.09.022. Epub 2014 Nov 4. PMID 25439600
- [Background] Tong AY, El-Dairi M, Maldonado RS, Rothman AL, Yuan EL, Stinnett SS, Kupper L, Cotten CM, Gustafson KE, Goldstein RF, Freedman SF, Toth CA. Evaluation of optic nerve development in preterm and term infants using handheld spectral-domain optical coherence tomography. Ophthalmology. 2014 Sep;121(9):1818-26. doi: 10.1016/j.ophtha.2014.03.020. Epub 2014 May 6. PMID 24811961
- [Background] Rothman AL, Folgar FA, Tong AY, Toth CA. Spectral domain optical coherence tomography characterization of pediatric epiretinal membranes. Retina. 2014 Jul;34(7):1323-34. doi: 10.1097/IAE.0000000000000113. PMID 24691567
- [Background] Maldonado RS, Yuan E, Tran-Viet D, Rothman AL, Tong AY, Wallace DK, Freedman SF, Toth CA. Three-dimensional assessment of vascular and perivascular characteristics in subjects with retinopathy of prematurity. Ophthalmology. 2014 Jun;121(6):1289-96. doi: 10.1016/j.ophtha.2013.12.004. Epub 2014 Jan 21. PMID 24461542
- [Background] Gramatikov BI, Irsch K, Guyton D. Optimal timing of retinal scanning during dark adaptation, in the presence of fixation on a target: the role of pupil size dynamics. J Biomed Opt. 2014;19(10):106014. doi: 10.1117/1.JBO.19.10.106014. PMID 25349032
- [Background] Irsch K, Gramatikov BI, Wu YK, Guyton DL. Improved eye-fixation detection using polarization-modulated retinal birefringence scanning, immune to corneal birefringence. Opt Express. 2014 Apr 7;22(7):7972-88. doi: 10.1364/OE.22.007972. PMID 24718173
- [Background] Gramatikov BI. Modern technologies for retinal scanning and imaging: an introduction for the biomedical engineer. Biomed Eng Online. 2014 Apr 29;13:52. doi: 10.1186/1475-925X-13-52. PMID 24779618
- [Background] Carrasco-Zevallos OM, Qian R, Gahm N, Migacz J, Toth CA, Izatt JA. Long working distance OCT with a compact 2f retinal scanning configuration for pediatric imaging. Opt Lett. 2016 Nov 1;41(21):4891-4894. doi: 10.1364/OL.41.004891. PMID 27805643
- [Background] Qian R, Carrasco-Zevallos OM, Mangalesh S, Sarin N, Vajzovic L, Farsiu S, Izatt JA, Toth CA. Characterization of Long Working Distance Optical Coherence Tomography for Imaging of Pediatric Retinal Pathology. Transl Vis Sci Technol. 2017 Oct 16;6(5):12. doi: 10.1167/tvst.6.5.12. eCollection 2017 Oct. PMID 29057163